CLINICAL TRIAL: NCT03848806
Title: A Phase II Multicenter Randomized Double-blind Comparator-Controlled Trial of HAT1 Compared to Calcipotriol in Patients With Mild to Moderate Chronic Plaque Psoriasis
Brief Title: Efficacy and Safety of HAT1 Compared to Calcipotriol in Patients With Mild to Moderate Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haus Bioceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCTP15MDZ1
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — calcipotriene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAT1 topical (Experimental): HAT1 topical cream will come in a blinded bottle. Patients, investigators, and the trial sponsor will be unaware of the trial group assignments. Packaging and labeling of the test and comparator products will be identical to maintain the blind.
  Interventions: Drug: HAT1
- Calcipotriol (Active Comparator): Calcipotriol topical cream will come in a blinded bottle. Patients, investigators, and the trial sponsor will be unaware of the trial group assignments. Packaging and labeling of the test and comparator products will be identical to maintain the blind.
  Interventions: Drug: Calcipotriol

INTERVENTIONS:
Drug: HAT1 — During the treatment phase, patients will be ask to apply the product twice daily on all lesional areas. The research team will provide instructions for the correct application of the treatment. If a lesion disappears, patients will continue applying the cream twice daily to the area. No additional creams, lotions or soaps other than provided test products will be allowed throughout the duration of the study.
  Arms: HAT1 topical
Drug: Calcipotriol — During the treatment phase, patients will be ask to apply the product twice daily on all lesional areas. The research team will provide instructions for the correct application of the treatment. If a lesion disappears, patients will continue applying the cream twice daily to the area. No additional creams, lotions or soaps other than provided test products will be allowed throughout the duration of the study.
  Other Names: Calcipotriol 0.005%
  Arms: Calcipotriol

SUMMARY:
Psoriasis, the most prevalent autoimmune disease in the U.S., manifests with plaque type psoriasis vulgaris with lesions localized to the scalp, postauricular region, face, diaper area, elbows, and knees. Inadequately controlled disease is common and a significant cause of extensive psychological and clinical morbidity in children. In addition, the safety and tolerability issues of common treatments for psoriasis including topical corticosteroids, calcipotriol, oral cytotoxic drugs, and biologic agents are especially problematic in patients that limit their use. Identification of therapies with high efficacy and safety profiles suitable for patients with psoriasis is therefore an area of critical unmet need. Haus Bioceuticals has developed a topical treatment for psoriasis denoted HAT1 (based on ingredients that have established clinical benefit), and have demonstrated that HAT1 is safe and profoundly effective in the treatment of psoriasis. This study is aimed to further evaluate the efficacy and safety of HAT1 compared to commonly used calcipotriol in patients with mild to moderate chronic plaque psoriasis.

DETAILED DESCRIPTION:
This is a randomized, double-blind trial. All patients who meet entry criteria will be randomized to receive either topical HAT01 or calcipotriol to be applied to the affected area 2 times per day. Treatment will continue for a maximum of 12 weeks. During all study visits, patients will be evaluated for efficacy and safety. The study will comprise of a 1 week washout period. During the washout period, patients will be asked to avoid using any products on their body including topical corticosteroids, ointments, creams, etc. During the treatment phase, patients will be provided one of the two test products to use twice daily on all lesional areas. No additional ointments or creams will be allowed throughout the duration of the study. Measurements and assessments will be taken according to the schedule. Patients will be followed through 12 weeks till the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of active plaque psoriasis with a minimum PGA score of 2 but not greater than 4
* Males or Females between 12-60 years
* Treatment area amenable to topical treatment
* Attending a hospital outpatient clinic or the private practice of a dermatologist
* Following verbal and written information about the trial, the patient must provide signed and dated informed consent before any study related activity is carried out, including activities relating to washout period.

Exclusion Criteria:

* Currently have non-plaque forms of psoriasis, eg, erythrodermic, guttate, or pustular psoriasis or a drug induced form of psoriasis.
* Systemic treatment with immunosuppressive drugs or corticosteroids within 4 weeks prior to enrollment. (Inhaled or intranasal steroids for asthma or rhinitis may be used)
* Topical treatment with immunomodulators or corticosteroids within 4 weeks prior to enrollment.
* Phototherapy treatment within 4 weeks prior to enrollment.
* Other topical therapy on the treatment area within 1 week prior to enrollment.
* Use of anti-histamine treatment during the study
* Clinical infection on the treatment area.
* Patients with history of cancer including skin cancer.
* Patients with history of an immunocompromised disease.
* Current participation in any other interventional clinical trial.
* Pregnancy or risk of pregnancy, and/or lactation
* History of allergy of any herbal components in HAT1
* Subjects with intense sun exposure during the study
* Patients known or suspected of not being able to comply with a trial protocol (e.g. alcoholism, drug dependency, or psychotic state)

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 174 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2016-09-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who achieve a Psoriasis Area and Severity Index (PASI) 75 response | Time Frame: Baseline to week 12
  75% or greater reduction from baseline in the PASI score

SECONDARY OUTCOMES:
Percentage of patients who achieve a Psoriasis Area and Severity Index (PASI) 50 response | Time Frame: Baseline to week 12
  50% or greater reduction from baseline in the PASI score
Percentage of patients achieving a Physicians Global Assessment (PGA) of Clear or Minimal at Week 12 | Time Frame: Baseline to week 12
  Reduction of PGA score from baseline to 0 (clear) or 1 (minimal disease)
Incidence of treatment emergent adverse events | Time Frame: Baseline to week 12
  Each patient were assessed for treatment emergent adverse events as part of safety assessments.